CLINICAL TRIAL: NCT06231706
Title: ZOE BIOME Study: Biotics Influence on Microbiome Ecosystem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Zoe Global Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BIOME
Record Dates: First submitted 2024-01-15; First posted 2024-01-30 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-05

CONDITIONS: Gut Microbiome; Prebiotic; Probiotic; Postprandial Period
Keywords: Gut Microbiome; Hunger; Mood; Energy; Postprandial
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Phase 1: Parallel arm randomised control trial Phase 2: Randomised crossover trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Phase 1: Control (Placebo Comparator): A commercially available bread crouton product. To be consumed as 2 x 14g portions per day for 6 weeks.
  Interventions: Other: Bread Crouton
- Phase 1: Intervention treatment (Experimental): Prebiotic-like nut and seed mix. To be consumed as 2 x 15g portions per day for 6 weeks
  Interventions: Other: Prebiotic-like nut and seed mix
- Phase 1: Secondary Intervention treatment. (Other): Probiotic capsule. To be consumed as one capsule per day for 6 weeks.
  Interventions: Dietary Supplement: Probiotic capsule
- Phase 2: Control (Placebo Comparator): Control breakfast consisting of White bread (3 slices; 128g approx.) and low fat spread (10-15g)
  Interventions: Other: White bread and low fat spread
- Phase 2: Intervention (Experimental): Intervention breakfast consisting of White bread (3 slices; 128g approx.) and low fat spread (10-15g) + Prebiotic-like nut and seed mix (2 x 15g portions)
  Interventions: Other: Prebiotic-like nut and seed mix; Other: White bread and low fat spread

INTERVENTIONS:
Other: Prebiotic-like nut and seed mix — A mixture of nuts, seeds and other plant based ingredients.
  Arms: Phase 1: Intervention treatment; Phase 2: Intervention
Other: Bread Crouton — A commercially available bread crouton product.
  Arms: Phase 1: Control
Dietary Supplement: Probiotic capsule — Contains the single strain Lactobacillus rhamnosus GG at 15 billion CFUs per capsule.
  Arms: Phase 1: Secondary Intervention treatment.
Other: White bread and low fat spread — Consists of 3 slices of bread (providing approx. 55-60g CHO; 3g fibre) + low fat spread (10-15g)
  Arms: Phase 2: Control; Phase 2: Intervention

SUMMARY:
The differences observed in host gut microbiome communities between health and disease states, and between different dietary patterns, has led to an increase in the use of dietary modulations to influence microbiome composition, both in research and in commercial contexts. Two particular groups of gut-active compounds include prebiotics (providing a direct source of nutrition that can stimulate host-beneficial microbiota as they are indigestible to the host) and probiotics (providing a direct source of live microorganisms that may potentially colonise the gut after reaching the large intestine, thus altering gut microbiome dynamics). Using a randomised controlled parallel trial design, the ZOE BIOME Study aims to investigate the efficacy of prebiotic and probiotic compounds in improving health outcomes including gut microbiome composition, gastrointestinal symptoms, and cardiometabolic markers of lipaemic, glycaemic and inflammatory status in a remote setting.

Further, consumption of high fibre supplements or food ingredients in combination with high carbohydrate meals has been shown to decrease the postprandial glycaemic response. To investigate the acute metabolic effects of prebiotic compounds , a randomised controlled crossover design postprandial study will be conducted. The ZOE BIOME Postprandial Study aims to investigate the efficacy of prebiotic compounds in improving acute postprandial glycaemic response, subjective feelings of hunger, satiety, mood, and subsequent eating behaviours.

DETAILED DESCRIPTION:
Phase 1:

A considerable body of evidence highlights the close association between the gut microbiome and health, with the roles performed by the microbiome spanning many functions. Firstly, intestinal microbiota are capable of digesting nutrients otherwise inaccessible to humans through gut physiology, to produce short-chain fatty acids, which are the primary energy source for intestinal epithelial cells. Secondly, the microbiome is part of the bi-directional relationship with host immunity and is involved in human immune homeostasis and immunological recognition that is both innate and adaptive. Moreover, dysbiosis of the gut microbiome has been reported in multiple disease states, including irritable bowel disease, inflammatory bowel disease, gut infections, cardiovascular disease, and psychological conditions such as depression and anxiety.

The differences observed in host gut microbiome communities between healthy and diseased states, and between different dietary patterns, has led to an increase in the use of dietary modulations in an attempt to influence microbiome composition, both in research and in commercial contexts. Two particular groups of gut-active compounds include prebiotics (providing a direct source of nutrition that stimulate host-beneficial microbiota as they are indigestible to the host) and probiotics (providing a direct source of live microorganisms that may potentially colonise the gut after reaching the large intestine, thus altering gut microbiome dynamics). Both compounds can be found naturally in foods; for example, many nuts and seeds contain prebiotic compounds such as fibre. Furthermore, foods can also be functionally modified to increase their content of prebiotics and probiotics. Finally, dietary supplementation with such compounds has also been shown to confer positive effects on health. However, the efficacy of dietary interventions involving supplementation in improving health in disease-free, free-living populations is not well understood.

The present study aims to investigate the efficacy of prebiotic and probiotic compounds in improving health, using a randomised parallel controlled trial design of 6-week intervention duration, in a healthy UK adult population, in a remote setting. The study design includes 2 treatments and a control: (i) a prebiotic-like nut and seed mix, consisting of whole-food ingredients high in plant polyphenolic compounds, fibre and micronutrients; (ii) a single-strain probiotic containing Lactobacillus rhamnosus GG, provided in capsule form; (iii) a bread crouton acting as a control (which can be used in a functionally equivalent application to the prebiotic).

Recruitment:

Participants will be recruited from within the ZOE Nutrition Product queue and ZOE mailing list to take part in this study. This queue, or waitlist, consists of individuals who have purchased the ZOE Nutrition Product but have not yet taken part in it. The ZOE mailing list consists of individuals who have registered interest in ZOE Health research studies and consented to be contacted in future. In addition, those that have consented to be contacted will be permitted to share the invitation to join the study with friends and family who may be interested in participating. Each potential participant will receive a study invitation via email, with a link to an online Participant Information Sheet, and will complete a two-step eligibility screening, before being given the option to consent to the study.

Study Design:

The study period requiring interaction of participants with the study staff will span a total of 9 weeks. The first 3 weeks of this period form the onboarding or run-in phase, during which participants will get detailed protocol instructions that they can discuss verbally with study staff. They will also provide their baseline measures during this time, in the week immediately prior to the commencement of their treatment.

The treatment phase will take the form of a 6-week randomised-controlled trial. Participants will be randomly assigned to one of three dietary intervention arms, which all contain commercially available products or products that are in the process of being brought to market:

1. Prebiotic-like nut and seed mix, designed by ZOE Ltd. Consumed as 2 x15g portions per day for 6 weeks.
2. Probiotic capsule containing the single strain Lactobacillus rhamnosus GG. Consumed as a single capsule portion (providing 15 billion CFUs) per day for 6 weeks.
3. Bread croutons. Consumed in portions of 10 croutons twice per day for 6 weeks (this portion is isocaloric to the nut and seed mix).

Participants will be instructed to consume the product of their allocated treatment arm in addition to their habitual diet. They will be asked to ensure their habitual diet remains unchanged throughout the study.

During the study, participants will be asked to complete the following tasks:

Dietary intake questionnaires. Dietary intake will be measured as both short-term intake and habitual intake. Short-term intake will be assessed through the 24 hr recall online tool 'Intake24', to be completed at three timepoints throughout the study (baseline (week 0); midpoint (week 4); and end of treatment (week 6)). Each timepoint will consist of 3 Intake24 records filled out on 3 days (2 weekdays + 1 weekend day). Habitual intake will be assessed through the PREDICT-Food Frequency Questionnaire (PREDICT-FFQ, a validated tool, in press), at one time point during the study (at screening, used as baseline).

Eating behaviour questionnaire. The participant's eating behaviour including eating window and diet patterns will be assessed at baseline (week 0), midpoint (week 4) and endpoint (week 6).

Health history questionnaire. This will be completed at baseline only, and will measure the baseline medical and health status of the participant.

Nutritional, general well-being and bowel symptom questionnaires. Hunger, mood, energy, skin quality, gastrointestinal symptoms and bowel habits will be measured by an online survey, at baseline and weekly throughout the study (7 timepoints in total).

Anthropometrics (weight, height, hip and waist circumference) will be self-reported through an online survey, at baseline (week 0) and endpoint (week 6).

Lifestyle questionnaires. Sleep quality, sleep quantity, and level of physical activity will be assessed at baseline and weekly throughout the study (7 timepoints in total).

Participant adherence questionnaires. These will be used to confirm the quantity of the treatment product that has been consumed by the participant, and to measure self-reported participant compliance to the study tasks. This will be completed weekly throughout the study treatment phase (6 timepoints in total).

Stool sampling. Using an at-home sampling kit, participants will collect a stool sample at two points throughout the study (baseline (week 0) and endpoint (week 6)).

Finger-prick dried blood spot (DBS) tests. Participants will complete these using an at-home sampling kit, at two points throughout the study (baseline (week 0) and endpoint (week 6))

Communication with Study Staff:

All procedures involved in the trial will be performed remotely. Participants will complete a live welcome call with study staff via video call in order to brief participant on their allocated intervention and study procedures. Throughout the trial participants will have access to live communication with members of study staff via email and phone.

Phase 2:

Consumption of high fibre supplements or food ingredients in combination with high carbohydrate meals has been shown to decrease the postprandial glycaemic response. To investigate the acute health effects of the prebiotic-like nut and seed mix, on postprandial responses, a randomised controlled crossover design postprandial study will be conducted.

We hypothesise that consumption of a high carbohydrate breakfast in combination with the prebiotic-like nut and seed mix (2 x 15g portions = 9g fibre) will decrease the postprandial glycaemic response, and improve postprandial subjective ratings of hunger, mood and alertness in comparison to the consumption of a high carbohydrate breakfast alone (control). The impact of the nut and seed mix on subsequent eating behaviours (time to next meal, amount consumed at next meal) will be investigated. Using a randomised crossover design, the ZOE BIOME Postprandial Study aims to investigate the efficacy of prebiotic compounds in improving acute postprandial glycaemic response, subjective feelings of hunger, satiety, mood, and subsequent eating behaviours.

Trial Objectives:

The primary objective of the randomised crossover trial is to evaluate the efficacy of a prebiotic-like nut and seed mix in modulating acute postprandial glucose responses when co-ingested with a carbohydrate rich breakfast.

Recruitment:

Phase 2 will be completed in a sub-group of participants recruited to Phase 1 of this study. Participants who were randomised to the control arm, and have completed phase 1 of the BIOME study will be given the option to take part in Phase 2. Each potential participant will receive a study invitation via email, with a link to an online Participant Information Sheet, and will complete a two-step eligibility screening, before being given the option to consent to the study.

Design:

A randomised crossover trial design, in a healthy UK adult population. Participants will consume 2 test meals in duplicate in a random order. Each meal will be separated by a minimum 2 day washout period. Participants will consume control and test breakfast meals in duplicate and the postprandial glucose responses will be measured using data collected from continuous interstitial glucose monitors. Breakfast test meals will consist of commercially available food products (bread and low-fat spread) and a novel blend of whole-food ingredients high in plant polyphenolic compounds, fibre and micronutrients (prebiotic-like nut and seed mix). Following an overnight fast, participants will consume one of two test meals:

White bread (providing approx. 55-60g CHO; 3g fibre) + Low-fat spread (10-15g) + Prebiotic-like nut and seed mix (2 x 15g portions, ~9g Fibre).

White bread (providing approx. 55-60g CHO; 3g fibre) + Low-fat spread (10-15g)

Following consumption of the test meals participants will be asked to fast for 3 hours during which time they may only consume water (the amount of which will be recorded on the first test day and replicated across all test days).

During testing days participants will be asked to complete visual analog scales (VAS) regarding subjective levels of hunger and mood.

All procedures involved in the trial will be performed remotely. Participants will complete a live welcome call with study staff via video call in order to brief participants on the study procedures. Throughout the trial participants will have access to live communication with members of study staff via email and phone.

ELIGIBILITY:
Inclusion Criteria:

* Can provide written informed consent through an electronic consent form
* Are able and willing to comply to the study protocol
* Are willing to complete their study tasks on specified dates (including over the Easter Holidays)
* Have completed the PREDICT Food Frequency Questionnaire sent to them via email
* Have not completed the ZOE Nutrition product before
* Are willing to do any of the three treatments to which they may be allocated, and able to complete them safely
* Have BMI between 18.5 kg/m2 and 40 kg/m2
* Are any sex
* Are aged between 35 and 65 years old
* Are based in the UK for the duration of the study and can have a study kit delivered to their location

Exclusion Criteria:

* Cannot eat the test treatments safely and comfortably (suffer from inflammatory bowel disease, coeliac disease, Crohn's disease, irritable bowel syndrome, allergies or intolerances, chronic constipation or chronic diarrhoea)
* Have BMI of less than 18.5 kg/m2 or more than 40 kg/m2
* Follow a non-omnivore diet (vegan, vegetarian)
* Have high fermented food intake at baseline for the preceding month (≥7 servings per week)
* Have high fibre intake at baseline for the preceding month (≥20g per day)
* Taking medication or products in the last 3 months that may modify the measured study outcomes (Antibiotics, non-topical steroids or other immunosuppressive medicines, biologics, probiotics/prebiotics, metformin, chronic use of non-steroidal anti-inflammatory drugs)
* Have used opiate pain medicine for 8 or more days during the last 3 months
* Have used a proton pump inhibitor for 8 or more days during the last 3 months
* Are currently a smoker
* Have experienced a heart attack, stroke, or major surgery in last 2 months
* Have received treatment for cancer in the last 3 months
* Are currently pregnant, breastfeeding or planning a pregnancy
* Are suffering from eating disorders, type 1 or type 2 diabetes mellitus.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Phase 1: Microbiome Composition | Baseline and 6 weeks
  The change in relative abundance of microbiome species from baseline to endpoint, derived from metagenomic analysis of stool samples.
Phase 2: Peak postprandial interstitial glucose concentration (C-Max) | Within 3 hours post test meal consumption
  Difference in C-Max between intervention and control meals.

SECONDARY OUTCOMES:
Phase 1: Lipid blood profile | Baseline and 6 weeks
  The change in lipid markers (triglycerides, total cholesterol, HDL-C, LDL-C, and lipoproteins) from baseline to endpoint, measured through finger-prick dried blood spot samples analysed by metabolomics.
Phase 1: Hemoglobin A1C | Baseline and 6 weeks
  The change in Hemoglobin A1C (HbA1c) from baseline to endpoint, measured through finger-prick dried blood spot samples.
Phase 1: Inflammation | Baseline and 6 weeks
  The change in glycoprotein acetylation (GlycA) from baseline to endpoint, measured through finger-prick dried blood spot samples analysed by metabolomics.
Phase 1: Gastrointestinal symptoms | Baseline and 6 weeks
  The change in gastrointestinal symptoms throughout the study duration, measured through questionnaires administered online. Symptoms measured include abdominal bloating, bowel movement frequency and form, indigestion and others.
Phase 1: Hunger level | Baseline and 6 weeks
  The change in hunger level throughout the study duration, measured through questionnaires administered online.
Phase 1: Energy level | Baseline and 6 weeks
  The change in energy level throughout the study duration, measured through questionnaires administered online.
Phase 1: Mood | Baseline and 6 weeks
  The change in mood throughout the study duration, measured through questionnaires administered online.
Phase 1: Body weight | Baseline and 6 weeks
  The change in weight from baseline to endpoint, measured through questionnaires administered online.
Phase 1: Waist circumference | Baseline and 6 weeks
  The change in waist circumference from baseline to endpoint, measured through questionnaires administered online.
Phase 1: Sleep | Baseline and 6 weeks
  The change in sleep quantity and quality throughout the study duration, measured through questionnaires administered online.
Phase 1: Skin quality | Baseline and 6 weeks
  The change in skin quality throughout the study duration, measured through questionnaires administered online.
Phase 2: Postprandial interstitial glucose (2h iAUC) | 2 hours post test meal consumption
  Difference in 2h iAUC between intervention and control test meals measured using continuous interstitial glucose monitors.
Phase 2: Postprandial Interstitial Glucose Time to Max Concentration (T-Max) | Within 3 hours post test meal consumption
  Difference in T-Max between intervention and control test meals measured using continuous interstitial glucose monitors.
Phase 2: Postprandial Interstitial Glucose dips (2-3h dips) | 2-3 hours post test meal consumption
  Difference in 2-3h dips between intervention and control test meals measured using continuous interstitial glucose monitors.
Phase 2: Postprandial Glucose (time course) | 3 hours post test meal consumption.
  Difference in time course responses of postprandial glucose between intervention and control test meals measured using continuous interstitial glucose monitors.
Phase 2: Postprandial subjective ratings of hunger (3h iAUC) | 3 hours post test meal consumption.
  Difference in iAUC between intervention and control test meals assessed using visual analog scales.
Phase 2: Postprandial subjective ratings of hunger (time-course) | 3 hours post test meal consumption
  Difference in time course responses of postprandial hunger between intervention and control test meals assessed using visual analog scales.
Phase 2: Postprandial subjective ratings of mood (3h iAUC) | 3 hours post test meal consumption.
  Difference in iAUC between intervention and control test meals assessed by visual analog scales.
Postprandial subjective ratings of Mood (time course) | 3 hours post test meal consumption
  Difference in time course responses of postprandial mood between intervention and control test meals assessed by visual analog scales.
Phase 2: Time to next meal | Anticipated 3-6 hours post test meal consumption
  Difference in time taken to consume next meal between intervention and control test meals assessed by physical food diary.
Phase 2: Amount Consumed at Next Meal | Anticipated 3-6 hours post test meal consumption
  Difference in amount consumed next meal between intervention and control test meals assessed by physical food diary.
Phase 2: Nutrient intake at the next meal | Anticipated 3-6 hours post test meal consumption
  Difference in nutrient intake at next meal between intervention and control test meals assessed by physical food diary.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Berry, Dr, Principal Investigator — King's College London, ZOE Ltd; Tim Spector, Pr, Principal Investigator — King's College London, ZOE Ltd
Locations (1):
- King's College London, London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flint HJ, Duncan SH, Scott KP, Louis P. Links between diet, gut microbiota composition and gut metabolism. Proc Nutr Soc. 2015 Feb;74(1):13-22. doi: 10.1017/S0029665114001463. Epub 2014 Sep 30. PMID 25268552
- [Background] Morrison DJ, Preston T. Formation of short chain fatty acids by the gut microbiota and their impact on human metabolism. Gut Microbes. 2016 May 3;7(3):189-200. doi: 10.1080/19490976.2015.1134082. Epub 2016 Mar 10. PMID 26963409
- [Background] Shreiner AB, Kao JY, Young VB. The gut microbiome in health and in disease. Curr Opin Gastroenterol. 2015 Jan;31(1):69-75. doi: 10.1097/MOG.0000000000000139. PMID 25394236
- [Background] Tang WH, Wang Z, Levison BS, Koeth RA, Britt EB, Fu X, Wu Y, Hazen SL. Intestinal microbial metabolism of phosphatidylcholine and cardiovascular risk. N Engl J Med. 2013 Apr 25;368(17):1575-84. doi: 10.1056/NEJMoa1109400. PMID 23614584
- [Background] Andrioaie IM, Duhaniuc A, Nastase EV, Iancu LS, Lunca C, Trofin F, Anton-Paduraru DT, Dorneanu OS. The Role of the Gut Microbiome in Psychiatric Disorders. Microorganisms. 2022 Dec 9;10(12):2436. doi: 10.3390/microorganisms10122436. PMID 36557689
- [Background] Peng M, Tabashsum Z, Anderson M, Truong A, Houser AK, Padilla J, Akmel A, Bhatti J, Rahaman SO, Biswas D. Effectiveness of probiotics, prebiotics, and prebiotic-like components in common functional foods. Compr Rev Food Sci Food Saf. 2020 Jul;19(4):1908-1933. doi: 10.1111/1541-4337.12565. Epub 2020 May 26. PMID 33337097
- [Background] Ballini A, Santacroce L, Cantore S, Bottalico L, Dipalma G, Vito D, Saini R, Inchingolo F. Probiotics Improve Urogenital Health in Women. Open Access Maced J Med Sci. 2018 Oct 20;6(10):1845-1850. doi: 10.3889/oamjms.2018.406. eCollection 2018 Oct 25. PMID 30455760
- [Background] Jenkins AL, Kacinik V, Lyon M, Wolever TM. Effect of adding the novel fiber, PGX(R), to commonly consumed foods on glycemic response, glycemic index and GRIP: a simple and effective strategy for reducing post prandial blood glucose levels--a randomized, controlled trial. Nutr J. 2010 Nov 22;9:58. doi: 10.1186/1475-2891-9-58. PMID 21092221
- [Background] Chen CO, Rasmussen H, Kamil A, Du P, Blumberg JB. Orange Pomace Improves Postprandial Glycemic Responses: An Acute, Randomized, Placebo-Controlled, Double-Blind, Crossover Trial in Overweight Men. Nutrients. 2017 Feb 13;9(2):130. doi: 10.3390/nu9020130. PMID 28208806